CLINICAL TRIAL: NCT05815784
Title: Myopia Control in the Pediatric Population: a Comparison of MiSight, Naturalvue Multifocal, and Atropine 0.05%
Brief Title: Myopia Control: a Comparison Study Between Atropine and MiSight
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Ann & Robert H Lurie Children's Hospital of Chicago (Other)
Responsible Party: Principal Investigator, Magdalena Stec, Assistant Professor of Ophthalmology, Ann & Robert H Lurie Children's Hospital of Chicago
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2022-5570
Record Dates: First submitted 2023-03-08; First posted 2023-04-18 (Actual); Last update posted 2024-11-19 (Actual); Status verified 2024-11

CONDITIONS: Myopia
MeSH Terms: conditions — Myopia | interventions — Atropine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

ARMS (3):
- Observation (No Intervention): No treatment.
- Atropine (Other): 0.05% atropine. One drop per eye per day for 2 years.
  Interventions: Drug: Atropine
- MiSight contact lenses (Other): MiSight contact lenses. Daily wear for 2 years.
  Interventions: Device: MiSight contact lenses

INTERVENTIONS:
Drug: Atropine — 0.05% atropine. One drop per eye per day for 2 years.
  Arms: Atropine
Device: MiSight contact lenses — Daily wear for 2 years.
  Arms: MiSight contact lenses

SUMMARY:
This research project aims to provide additional knowledge of pharmacological and optical methods of myopia control and to gain a better understanding of the biometry of the pediatric eye, which contributes to the onset and progression of myopia. As a result, this study will improving our best practices for myopia control in pediatric patients.

ELIGIBILITY:
Inclusion Criteria:

* Children age of 5-12 years old at their baseline exam
* Children with a spherical equivalent refractive error of +0.50D (minimal hyperopia) to -7.50 D (high myopia)
* Gestational age ≥ 32 weeks.
* Birth weight >1500g.

Exclusion Criteria:

* Current or previous form of myopia control
* Current or previous use of bifocal, progressive- addition lenses, or multifocal contact lenses
* Known atropine allergy or contact lens intolerance (allergy to only one can still allow enrollment in the other group)
* Abnormality of cornea, lens, central retina, iris, or ciliary body
* Current or prior history of manifest strabismus, amblyopia, or nystagmus
* Current or previous myopia treatment with atropine, pirenzepine or another anti-muscarinic agent.
* Current or previous use of bifocals, progressive-addition lenses, or multi-focal contact lenses.
* Current or previous use of orthoK, rigid gas permeable, or other contact lenses being used to reduce myopia progression.
* Abnormality of the cornea, lens, central retina, iris, or ciliary body.
* Prior eyelid, strabismus, intraocular, or refractive surgery.
* Down syndrome or cerebral palsy.
* Diseases known to affect accommodation, vergence, or ocular motility (e.g., multiple sclerosis, Grave's disease, myasthenia gravis, diabetes mellitus, Parkinson's disease)
* Existing ocular conditions (e.g., retinal disease, cataracts, ptosis) or systemic/neurodevelopmental conditions (e.g., Down syndrome) which may influence refractive development
* Any condition that in the judgement of the investigator could potentially influence refractive development.
* Existing conditions that may affect the long-term health of the eye or require regular pharmacologic treatment that may adversely interact with study medication (e.g., JIA, glaucoma, diabetes mellitus, pre-diabetes)
* Inability to comprehend and/or perform any study-related clinical tests

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 348 (Estimated)
Dates: Start 2023-05-02 (Actual); Primary Completion 2026-03-13 (Estimated); Study Completion 2026-03-13 (Estimated)

PRIMARY OUTCOMES:
axial length | 2 years
  change in axial length (as measured by biometry) over a 2-year time period
Refractive error | 2 years
  change in refractive error over a 2-year time period

SECONDARY OUTCOMES:
compliance with treatment | 2 years
reported side effects | 2 years
success rate of contact lens fitting in the younger children | 2 years
contact lens tolerance in the younger children | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Magdalena Stec, OD, Principal Investigator — Ann & Robert H Lurie Children's Hospital of Chicago
Locations (1):
- Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois, United States